CLINICAL TRIAL: NCT03564847
Title: Testing Low-cost Learning Through Play (LTP) Plus Parenting Intervention for Depressed Fathers (LTP Plus Dads) A Cluster Randomized Controlled Trial (RCT)
Brief Title: Learning Through Play (LTP) Plus Intervention for Depressed Fathers (LTP Plus Dads)
Acronym: LTP+Dads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Grand Challenges Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-LTP Plus Dads-002
Record Dates: First submitted 2018-05-23; First posted 2018-06-21 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Depression
Keywords: Learning Through Play Plus; Cognitive Behavior Therapy; Parenting Intervention; Low and middle-income country
MeSH Terms: conditions — Depression | interventions — Long-Term Potentiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers doing outcome assessment will be kept blind to the group allocations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP Plus (Experimental): LTP Plus Participants will receive the intervention over 4 months Weekly sessions for 2 months and fortnightly for next two months by trained non-specialists/community health workers.
  Interventions: Behavioral: LTP Plus
- Treatment As Usual (TAU) (No Intervention): Treatment as Usual (TAU) group will receive routine care and their follow up will be done at 4th and 6th month post randomization.

INTERVENTIONS:
Behavioral: LTP Plus — LTP+Dads is a 12 - session group integrated parenting intervention: i.e LTP (Learning through Play) which includes a pictorial calendar, consisting of stages of child development from birth to 3 years. It includes parent-child play and other activities that promote parental involvement, learning, and attachment. In each stage, there are five areas of child development: sense of self, physical, relationships, understanding, and communication. All areas are written in simple, low-literacy language.
  Second component of intervention is CBT adapted from Jeanne Miranda manual (Group CBT for Depression, group leaders guide book-2006) focusing on the three areas: thoughts and your mood, activities and your mood, people interaction and your mood.
  Third component of intervention is content taken from Ed Bader's manual (Focus on Fathers) includes importance of fathers in child development, stress management at work and home, budgeting, anger management, conflict resolution and time management.
  Arms: LTP Plus

SUMMARY:
The aim of the study is to evaluate the clinical and cost effectiveness of culturally adapted group parenting intervention delivered by non-specialists and community health workers for depressed fathers.

DETAILED DESCRIPTION:
Most research on the association between parental depression and child outcomes has focused mainly on mothers. However, studies suggest that the relationship between parental depression and child outcome is not necessarily limited to mothers.

The study has two phases quantitative and qualitative:

Purpose of this quantitative phase is to determine if the LTP plus programme delivered by non-specialists and community health workers reduces symptoms of paternal depression and improves child development compared to treatment as usual.

In the qualitative part of the study focus groups and in-depth digitally recorded interviews will be conducted with participants by trained research staff at two-time points both before and after the intervention. These focus groups and in-depth interviews will continue till the data saturation is achieved. In addition, Participants who refused to participate in the trial will be asked if they would be willing to be contacted by a researcher to discuss their reasons for not taking part. Moreover, in-depth digitally-recorded interviews with stakeholders (grandparents, therapists, health professionals, etc) will also be conducted by trained researchers.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years old fathers
* Having children aged between 0-30 months
* Diagnosis of major depressive disorder using the Structure Clinical Interview for DSM-V,
* Ability to complete a baseline assessment.
* Given written informed consent

Exclusion Criteria:

* Any medical illness that will prevent them from participation in the clinical trial,
* Current or past diagnosis of bipolar depression
* Currently using antidepressants or receiving any kind of psychotherapy
* Active suicidal ideation,
* Any other severe physical or mental disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only Fathers will be included in the study
Enrollment: 357 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale HAM-D 17 (Hamilton, 1960) | Changes from Baseline to 4th and 6th Month
  The questionnaire is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. The HAM-D is a simple 17 item self-report questionnaire can also be administered by a trained research worker. The translated version of the scale has been used in previous studies in Pakistan (Husain et al., 2017). It takes about 10 to 15 minutes to administer this scale. A score of 0-7 indicates normal, 8-13 mild depression, 14-18 moderate depression, 19-22 severe depression and > 22 severe depression

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD) 7 (Spitzer, Kroenke, Williams, & Löwe, 2006): | Changes from Baseline to 4th and 6th Month
  The GAD-7 is a 7-item scale used to screen for and measure severity of generalized anxiety disorder. Scores of 5, 10 & 15 are taken as cut-off points for mild, moderate and high. it takes about 5 minutes to administer this scale.
Rosenberg's Self-Esteem Scale (Rosenberg, 1995) | Changes from Baseline to 4th and 6th Month
  Rosenberg's Self-Esteem Scale will be used to measure self-esteem and personal worthlessness. It is a simple 9 item questionnaire. Higher scores indicate higher self-esteem. The Urdu translated version of scale has been used in our previous studies in Pakistan. (Husain et al 2014; Husain et al., 2017).The scale takes about 5 to 10 minutes to administer
Brief Disability Questionnaire BDQ:(Von Korff, Ustun, Ormel, Kaplan, & Simon, 1996) | Changes from Baseline to 4th and 6th Month
  BDQ is a simple 8 Items questionnaire to measure disability in the physical or social life. Total scores across items 1-6 are considered to indicate 'moderate' and 'severe' disability for score ranges 8-13 and 14-22 respectively. The translated version of scale has been used in previous trials in Pakistan (Naeem et al., 2015). It takes about 5 to 10 minutes to administer this scale
Patient Health Questionnaire (PHQ-9) (Kroenke, Spitzer, & Williams, 2003) | Changes from Baseline to 4th and 6th Month
  The Patient health Questionnaire (PHQ-9) is 10 items self-report questionnaire which is easy to use and can be administered by a trained research worker. Score ranges from : 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe
Client Satisfaction Questionnaire (CSQ) (Attkisson & Greenfield, 1995) | After completion of the intervention at 4th month only
  The participants will rate their satisfaction with the intervention at 4th month using the CSQ, it comprises of 8 items, high scores indicate greater satisfaction (Attkisson & Greenfield, 1995). it takes about 5 minutes to administer this scale
Parenting Scale (Arnold, O'leary, Wolff, & Acker, 1993) | Changes from Baseline to 4th and 6th Month
  Parent-completed 30-item questionnaire measuring three dysfunctional discipline styles: (1) laxness (permissive discipline), (2) over-reactivity (authoritarian discipline) and (3) verbosity (reliance on talking), with responses rated on a seven-point scale. it takes about 10 minutes to administer this scale.
Euro-Qol-5 Dimensions (EQ-5D) ( Brooks R. EuroQol,.1996) | Changes from Baseline to 4th and 6th Month
  Health-related quality of life will be measured by using EQ-5D. This is a standardized instrument that measures five health dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each scored from 1 to 3 indicating "no problem" to "severe problems". In both the visual analogue scale, and the standardized valuation score, lower scores indicate poorer QOL. It takes about 5 minutes to administer this scale.
Hurt, Insulted, Threatened with Harm and Screamed (HITS) (Sherin, Sinacore, Li, Zitter, & Shakil, 1998): | Changes from Baseline to 4th and 6th Month
  HITS is simple 4 item domestic violence screening tool. Each item is scored from 1-5. Range between 4-20. A score greater than 10 signify that an individual are at risk of domestic violence. It takes about 5 minutes to administer this scale. An adapted version of the scale is being used in this study.
Dyadic Adjustment Scale (DAS):(Spanier, 1976) | Changes from Baseline to 4th and 6th Month
  DAS is a 32 items self-report questionnaire, to measure couple satisfaction and to assess how each partner perceives his/her relationship. The scale has good psychometric properties (Graham, Liu, & Jeziorski, 2006) and has also been used with depressed mothers (Wolman, Chalmers, Hofmeyr, & Nikodem, 1993). A total DAS score, ranging from 0 to 150, is derived by summing across the four subscales. The 32 items of the DAS are answered on Likert-type scales with questions representing each of the four subscales distributed throughout.It takes about 10 to 15 minutes to administer. The culturally adapted version of the scale is being used in this study.
Knowledge of Expectation and Child Development | Changes from Baseline to 4th and 6th Month
  A 25-item questionnaire will be used to assess paternal knowledge and expectations for child development in the first three years. Higher score indicated higher knowledge about child development. (Husain et al 2017) .It takes about 5 to 10 minutes to administer this scale
OSLO 3 (Nosikov & Gudex, 2003) | Changes from Baseline to 4th and 6th Month
  Oslo-3 Items social support scale focuses on the quality of social network, perceived positive interest and concern from other people and available help from neighbors if necessary. A score of 3-8 is "poor support", 9-11 is "moderate support" and 12-14 is "strong support". The Urdu version of the scale has already been used in previous studies in Pakistan(Husain, Chaudhry, Jafri, et al., 2014). it takes about 5 minutes to administer this scale.
Parenting Stress Index - Short Form (Abidin, 1995) | Changes from Baseline to 4th and 6th Month
  Parents rate 36 items on a five-point rating scale (1-5) on three sub scales: (1) Parenting Distress, (2) Difficult Child Characteristics, and (3) Dysfunctional Parent-Child Interaction. it takes about 10 to 15 minutes to administer this scale.
Eyberg Child Behaviour Inventory (ECBI) (Eyberg, Boggs, & Reynolds, 1980) | Changes from Baseline to 4th and 6th Month
  The ECBI is a parent rating scale consisting of items relating specifically to behaviors associated with conduct problems in children. The ECBI is a behaviorally specific instrument consisting of a list of 36 behaviors. It has two scales: (a) The Intensity Scale, which indicates how often these behaviors occur, and (b) The Problem Scale, identifying which specific behaviors are considered as problems by the parents. Rating on intensity scale will be done on seven-point (1-7) whereas on problem scale with YES or NO. it takes about 10-15 minutes to administer this scale.
Manchester Assessment of Caregiver-Infant Interaction (MACI) | Changes from Baseline to 6th Month
  It is designed as a global rating measure, covering general features of parents, infant and dyadic qualities of interaction. It comprises of seven rating scales that covers broad aspects of interaction between a primary caregiver and their infant, each with a seven point scale (Wan, Brooks, Green, Abel, & Elmadih, 2016). It is a method of systematically evaluating qualitative or global aspects of behavioural interaction between a primary caregiver and infant through rating their unstructured play from videotape. Ratings are made along a 7-point scale that show variance across the population Based on 6 minutes of caregiver-infant interaction videotaped in the lab or home.
Anthropometric measures (Weight) | Changes from Baseline, to 4th and 6th Month
  Weight will be measured in Kilograms
Anthropometric measures (Height) | Changes from Baseline, to 4th and 6th Month
  Height will be measured in centimeters
Anthropometric measures (Head Circumference) | Changes from Baseline, to 4th and 6th Month
  The measurement swill be taken with a device that cannot be stretched, such as a flexible metal tape measure.
Anthropometric measures (Arm Circumference) | Changes from Baseline, to 4th and 6th Month
  The measurement swill be taken with a device that cannot be stretched, such as a flexible metal tape measure.
Ages and Stages Social-Emotional Questionnaire(Squires et al., 2009) | Changes from Baseline to 4th and 6th Month
  This scale will be used to measure child development. Parents will report on their child's communication,gross motor, fine motor, problem solving and personal-social development. it takes about 10 minutes to administer this scale.
Infant development: Ages and Stages Questionnaire (Squires, Bricker, & Twombly, 2009) | Changes from Baseline to 4th and 6th Month
  This scale will be used to measure child development. Parents will report on their child's communication, gross motor, fine motor, problem solving and personal-social at different time points. it takes about 15 to 20 minutes to administer this scale
Bayley Scales of Infant Development (BSID-V3) (Bayley, Nancy (2006 | Changes from Baseline to 6th Month
  The Bayley Scales of Infant and Toddler Development is a standard series of measurements originally developed by psychologist Nancy Bayley used primarily to assess the development of infants and toddlers, ages 1-42 months. Scoring: 0 or 1 depending on if the child is able to perform the activity for cognitive, motor(fine and gross subscales), and language(expressive and receptive subscales) scored by examiner. Social-emotional and adaptive questionnaires filled out by parent/caregiver with same scale 0 or 1. The highest possible score on a subtest is 19, and the lowest possible score is 1. Scores from 8 to 12 are considered average.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhary, MD, Principal Investigator — PILL
Locations (2):
- Pakistan (2):
  - Bin Qasim Town, Karachi, Sindh
  - Orangi Town, Karachi, Sindh

REFERENCES:
- [Background] Hasin DS, Goodwin RD, Stinson FS, Grant BF. Epidemiology of major depressive disorder: results from the National Epidemiologic Survey on Alcoholism and Related Conditions. Arch Gen Psychiatry. 2005 Oct;62(10):1097-106. doi: 10.1001/archpsyc.62.10.1097. PMID 16203955
- [Background] Hirschfeld RM, Montgomery SA, Keller MB, Kasper S, Schatzberg AF, Moller HJ, Healy D, Baldwin D, Humble M, Versiani M, Montenegro R, Bourgeois M. Social functioning in depression: a review. J Clin Psychiatry. 2000 Apr;61(4):268-75. doi: 10.4088/jcp.v61n0405. PMID 10830147
- [Background] Husain MI, Chaudhry IB, Husain N, Khoso AB, Rahman RR, Hamirani MM, Hodsoll J, Qurashi I, Deakin JF, Young AH. Minocycline as an adjunct for treatment-resistant depressive symptoms: A pilot randomised placebo-controlled trial. J Psychopharmacol. 2017 Sep;31(9):1166-1175. doi: 10.1177/0269881117724352. Epub 2017 Aug 31. PMID 28857658
- [Background] Husain N, Chaudhry I, Raza-ur-Rehman, Ahmed GR. Self-esteem and obsessive compulsive disorder. J Pak Med Assoc. 2014 Jan;64(1):64-8. PMID 24605716
- [Background] Husain N, Chaudhry N, Jafri F, Tomenson B, Surhand I, Mirza I, Chaudhry IB. Prevalence and risk factors for psychological distress and functional disability in urban Pakistan. WHO South East Asia J Public Health. 2014 Apr-Jun;3(2):144-153. doi: 10.4103/2224-3151.206730. PMID 28607300
- [Background] Husain N, Parveen A, Husain M, Saeed Q, Jafri F, Rahman R, Tomenson B, Chaudhry IB. Prevalence and psychosocial correlates of perinatal depression: a cohort study from urban Pakistan. Arch Womens Ment Health. 2011 Oct;14(5):395-403. doi: 10.1007/s00737-011-0233-3. Epub 2011 Sep 4. PMID 21898171
- [Background] Kane P, Garber J. The relations among depression in fathers, children's psychopathology, and father-child conflict: a meta-analysis. Clin Psychol Rev. 2004 Jul;24(3):339-60. doi: 10.1016/j.cpr.2004.03.004. PMID 15245835
- [Background] Kaufman J, Yang BZ, Douglas-Palumberi H, Houshyar S, Lipschitz D, Krystal JH, Gelernter J. Social supports and serotonin transporter gene moderate depression in maltreated children. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17316-21. doi: 10.1073/pnas.0404376101. Epub 2004 Nov 24. PMID 15563601
- [Background] Klein DN, Lewinsohn PM, Rohde P, Seeley JR, Olino TM. Psychopathology in the adolescent and young adult offspring of a community sample of mothers and fathers with major depression. Psychol Med. 2005 Mar;35(3):353-65. doi: 10.1017/s0033291704003587. PMID 15841871
- [Background] Naeem F, Gul M, Irfan M, Munshi T, Asif A, Rashid S, Khan MN, Ghani S, Malik A, Aslam M, Farooq S, Husain N, Ayub M. Brief culturally adapted CBT (CaCBT) for depression: a randomized controlled trial from Pakistan. J Affect Disord. 2015 May 15;177:101-7. doi: 10.1016/j.jad.2015.02.012. Epub 2015 Feb 23. PMID 25766269
- [Background] Ramchandani P, Stein A, Evans J, O'Connor TG; ALSPAC study team. Paternal depression in the postnatal period and child development: a prospective population study. Lancet. 2005 Jun 25-Jul 1;365(9478):2201-5. doi: 10.1016/S0140-6736(05)66778-5. PMID 15978928
- [Derived] Husain MI, Kiran T, Sattar R, Khoso AB, Wan MW, Singla DR, Umer M, Mangrio R, Bassett P, Chaudhry IB, Zafar SN, Jafri FA, Chaudhry N, Husain N. A Group Parenting Intervention for Male Postpartum Depression: A Cluster Randomized Clinical Trial. JAMA Psychiatry. 2025 Jan 1;82(1):22-30. doi: 10.1001/jamapsychiatry.2024.2752. PMID 39356541